CLINICAL TRIAL: NCT05864716
Title: The Comparison of the Effect of Probiotics Between Delivery Via Colonoscopic Spray and Oral Administration in the Treatment of Irritable Bowel Syndrome
Brief Title: Colonoscopic Probiotics Spray in Irritable Bowel Syndrome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A BR 111 0 47
Record Dates: First submitted 2023-04-03; First posted 2023-05-18 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-04

CONDITIONS: Effect of Drug
Keywords: Irritable bowel syndrome; Probiotics; Colonoscopic spray
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Placebo powder was applied in the control group, and the powder was prepared in probiotics factory, which was blind to both patients and caregivers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- probiotics-spray (PS) group (Experimental): In the PS group, 1 vial of multi-strain probiotics powder via colonoscopic spray is performed once, followed by five-days of two oral placebo capsules daily. After the five-day treatment, the 2nd fecal sample will be collected. Both groups will receive a 23-day course of oral probiotics (two capsules twice daily) subsequently. The patients were asked to keep a diary to record bowel habits and register any adverse events. The 3rd fecal sample will be collected 28 days after the colonoscopy. The questionnaires will be completed 28 days and 84 days after the colonoscopy to assess responses of treatment. Polyethylene glycol and loperamide were allowed during the intervention as the rescue medication.
  Interventions: Biological: Colonscopic probiotics spray
- probiotics-oral (PO) group (Active Comparator): In the PO group, 1 vial of placebo powder via colonoscopic spray is performed once, followed by five-days of two oral probiotics capsules daily. After the five-day treatment, the 2nd fecal sample will be collected. Both groups will receive a 23-day course of oral probiotics (two capsules twice daily) subsequently. The patients were asked to keep a diary to record bowel habits and register any adverse events. The 3rd fecal sample will be collected 28 days after the colonoscopy. The questionnaires will be completed 28 days and 84 days after the colonoscopy to assess responses of treatment. Polyethylene glycol and loperamide were allowed during the intervention as the rescue medication.
  Interventions: Biological: Colonscopic probiotics spray

INTERVENTIONS:
Biological: Colonscopic probiotics spray — 20g of multi-strain probiotics powder via colonoscopic spray. The probiotic used in this study is SynPro-15G, which has 15 probiotics, including Bacillus coagulans BC1031, Bifidobacterium bifidum BB14, Bifidobacterium breve BR18, Bifidobacterium animalis subsp. lactis BAL06, Bifidobacterium longum (B. longum) BL986, Lactobacillus acidophilus LA1063, Lactobacillus casei LC122, Lactobacillus delbrueckii subsp. lactis LDL114, Lactobacillus fermentum LF26, Lactobacillus helveticus LH43, Lactobacillus paracasei LPC12, Lactobacillus plantarum LP198, Lactobacillus reuteri LR21, Lactobacillus rhamnosus LRH10, and Streptococcus thermophilus ST37 at a concentration of 2x1010 CFU/g (Synbiotech Corp., Kaohsiung, Taiwan). SynPro-15G is made either as a vial of powder (2x1011 CFU /vial) for colonoscopic spray or as a capsule (2x1010 CFU/capsule) for oral intake.

SUMMARY:
Irritable bowel syndrome (IBS) is a common chronic functional disorder of the gastrointestinal (GI) tract characterized by chronic abdominal pain and altered bowel habits without organic disease. IBS is associated with substantial costs to patients, healthcare system and society in terms of increased health care expenditures, loss of work productivity and decrease in quality of life (QoL). Multiple factors play an important role in the pathogenesis of IBS, including disturbed gut microbiota (dysbiosis). Fecal microbiota transplantation (FMT) and probiotics administration can manipulate the disturbed intestinal microbiota. According to previous studies, inconsistent efficacy of oral probiotic administration was reported. FMT may have good and lasting efficacy, but the donor selection and route of administration are still issues. Direct delivery of probiotics into the colon by colonoscopy can ensure sufficient microbiota distribution in the colon, so faster and better efficacy may be expected. Therefore, this study is aimed toward validating the efficacy and safety of the colonoscopic probiotics-spray in IBS treatment.

Patients diagnosed with irritable bowel syndrome by Rome IV criteria will be enrolled in this randomized double-blind double-dummy parallel controlled study. The enrolled patients will be randomly assigned to the probiotics-spray (PS) group and the probiotics-oral (PO) group, respectively. The patients in the PS group will receive colonoscopic spray of probiotics once followed by oral placebo for 5 days, while the patients in the PO group will receive colonoscopic spray of placebo once followed by oral probiotics divided into 5 days. Then all of the patients will take the same dose of oral probiotics until 4 weeks. This study will evaluate the efficacy between the PS group and the PO group. Moreover, this study will compare the difference in fecal microbiota changes and safety between these two groups.

DETAILED DESCRIPTION:
Irritable bowel syndrome (IBS) is a common chronic functional disorder of the gastrointestinal (GI) tract characterized by chronic abdominal pain and altered bowel habits without organic disease. The global prevalence of IBS in 2012 was estimated to be 11.2%. The overall incidence of IBS in Taiwan was 106.54 per 10000 population from 2012 to 2018, which is similar to the global prevalence. IBS is associated with substantial costs to patients, healthcare system and society in terms of increased health care expenditures, loss of work productivity and decrease in quality of life (QoL). There is no definite treatment for IBS, and current available treatments are mainly directed at symptom relief.

The cause of IBS is not yet known; however, multiple factors play an important role in the pathogenesis of IBS, such as disturbed gut microbiota (dysbiosis), altered enteroendocrine cells, previous infections, genetics and diet. Treatment guidelines recommend medications focused on IBS symptoms, diets low in fermentable types of oligosaccharides, and the use of probiotics. Probiotics are live microorganisms using in dietary as supplemental products. They have the beneficial effect on gut microenvironment, and may be an effective treatment for global symptoms and abdominal pain in IBS. Probiotics were defined as live microbial feed supplements that benefit the host by improving the intestinal microbial balance. The strains most frequently used as probiotics belong to the genera Bifidobacterium and Lactobacillus. Some probiotics have anti-inflammatory activity while others can modulate visceral hypersensitivity. However, inconsistent efficacy of probiotic administration was reported in the previous literature. Hod K, et al. conducted a double-blind, placebo-controlled study to assess the effect of a probiotic mixture on symptoms and inflammatory markers in women with diarrhea-predominant IBS, but they did not demonstrate superiority of probiotics over placebo. However, some meta-analysis revealed efficacy of probiotics for treatment of IBS. A meta-analysis published in 2020 concluded the RR of IBS symptoms improvement or response with probiotics treatment was 1.52, however, with high heterogeneity. The duration, dose and single or combination of probiotics vary and need to be further evaluated. A review of probiotics in IBS suggests that probiotic supplements have a delayed eﬀect in the improvement of IBS symptoms. Khodadoostan M, et al. conducted a trial to evaluate the effect of probiotic administration immediately and 1 month after colonoscopy in diarrhea-predominant IBS patients, which revealed the use of probiotics had the beneficial effect on IBS symptoms. Furthermore, it can be said that reductions in symptoms and pain in the two treatment groups were not significantly different, but after 6 months of treatment, the effect of probiotics in patients who immediately use it after colonoscopy was more visible and more stable. Niu HL, et al studied the efficacy and safety of probiotics in patients with irritable bowel syndrome based on 35 randomized controlled trials, which reveals supplementation with a multi-strain probiotic has greater potential to improve IBS symptoms than a single strain, and there is also a trend toward a beneficial effect of Bifidobacterium on global IBS symptoms and pain scores. Therefore, investigators propose a trial to evaluate the efficacy of the use of multi-strain probiotics including Bifidobacterium which is immediately used after colonoscopy for IBS treatment.

It is novel to conduct the study to compare the efficacy and safety of probiotics which are delivered directly via colonoscopy and oral administration. The amount of stool for FMT is 30 to 100 grams; thus, around 1012 to 1013 CFU bacteria will be transplanted in an FMT procedure. In this trial, the investigators will transplant 2x1011 CFU multi-strain probiotics into the colon via colonoscopic spray. Probiotics may be safer than FMT due to minimal risk of transmission of pathogenic organisms. It is also easier to prepare probiotics than feces from a superdonor. If it works, colonoscopic probiotics spray may replace FMT in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Moderate-to-severe IBS symptoms, as indicated by a score of ≥175 on the IBS Severity Scoring System (IBS-SSS).

Exclusion Criteria:

* Presence of immune deficiency or treatment with immune-modulating medication.
* Pregnant or lactating.
* Severe psychiatric disorder, or alcohol or drug abuse.
* Use of probiotics or treatment with antibiotics within 4 weeks prior to study entry.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
A change in the IBS-SSS total score of ≥50 points | 84 days
  The primary endpoint is a reduction in the IBS-SSS total score of ≥50 points .Abdominal symptoms are assessed on Day 0, Day 5, Day 28 and Day 84 using the IBS-SSS questionnaires. Patients whose total IBS- SSS score decreased by ≥50 points after the intervention are considered responders. A decrease of ≥175 points in the IBS- SSS total score considered to indicate significant clinical improvements.

SECONDARY OUTCOMES:
The preservation of probiotics following intervention | 28 days
  The investigators will evaluate the gut microbiota by fecal qPCR in the PS group and PO group, respectively, on Day 0, Day 5 and Day 28. The investigators will also compare the relative abundance of target probiotics between the two study groups, such as Lactobacillus acidophilus, Bifidobacterium bifidum, Streptococcus thermophilus, or others.
The change of fecal microbiota following intervention | 28 days
  The investigators will evaluate the gut microbiota by fecal qPCR in the PS group and PO group, respectively, on Day 0, Day 5 and Day 28. The investigators will compare the distribution of gut microbiota between D0, D5, and D28
A reduction in the Hospital Anxiety and Depression Scale (HADS) | 84 days
  Hospital Anxiety and Depression Scale (HADS) are also used to assess the presence of anxiety and depression. HADS scale will be recorded on day 0 and day 84.
A reduction in Fatigue Assessment Scale (FAS) | 84 days
  Fatigue is measured using the Fatigue Assessment Scale (FAS). A decrease of ≥4 points in the FAS score are considered to indicate significant clinical improvements. FAS will be recorded on day 0 and day 84.

IPD SHARING:
Plan to Share IPD: Yes
After study completed and paper accepted
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 10 years

REFERENCES:
- [Result] Lovell RM, Ford AC. Global prevalence of and risk factors for irritable bowel syndrome: a meta-analysis. Clin Gastroenterol Hepatol. 2012 Jul;10(7):712-721.e4. doi: 10.1016/j.cgh.2012.02.029. Epub 2012 Mar 15. PMID 22426087
- [Result] Lai YT, Chen CY, Bair MJ. Epidemiology, Clinical Features, and Prescribing Patterns of Irritable Bowel Syndrome in Taiwan. Front Pharmacol. 2021 Dec 9;12:788795. doi: 10.3389/fphar.2021.788795. eCollection 2021. PMID 34975485
- [Result] Gralnek IM, Hays RD, Kilbourne A, Naliboff B, Mayer EA. The impact of irritable bowel syndrome on health-related quality of life. Gastroenterology. 2000 Sep;119(3):654-60. doi: 10.1053/gast.2000.16484. PMID 10982758
- [Result] Canavan C, West J, Card T. Review article: the economic impact of the irritable bowel syndrome. Aliment Pharmacol Ther. 2014 Nov;40(9):1023-34. doi: 10.1111/apt.12938. Epub 2014 Sep 9. PMID 25199904
- [Result] El-Salhy M. Recent advances in the diagnosis of irritable bowel syndrome. Expert Rev Gastroenterol Hepatol. 2015;9(9):1161-74. doi: 10.1586/17474124.2015.1067138. Epub 2015 Jul 15. PMID 26162959
- [Result] Mazzawi T. Gut Microbiota Manipulation in Irritable Bowel Syndrome. Microorganisms. 2022 Jun 30;10(7):1332. doi: 10.3390/microorganisms10071332. PMID 35889051
- [Result] Vasant DH, Paine PA, Black CJ, Houghton LA, Everitt HA, Corsetti M, Agrawal A, Aziz I, Farmer AD, Eugenicos MP, Moss-Morris R, Yiannakou Y, Ford AC. British Society of Gastroenterology guidelines on the management of irritable bowel syndrome. Gut. 2021 Jul;70(7):1214-1240. doi: 10.1136/gutjnl-2021-324598. Epub 2021 Apr 26. PMID 33903147
- [Result] Verdu EF, Bercik P, Verma-Gandhu M, Huang XX, Blennerhassett P, Jackson W, Mao Y, Wang L, Rochat F, Collins SM. Specific probiotic therapy attenuates antibiotic induced visceral hypersensitivity in mice. Gut. 2006 Feb;55(2):182-90. doi: 10.1136/gut.2005.066100. Epub 2005 Aug 16. PMID 16105890
- [Result] Hod K, Sperber AD, Ron Y, Boaz M, Dickman R, Berliner S, Halpern Z, Maharshak N, Dekel R. A double-blind, placebo-controlled study to assess the effect of a probiotic mixture on symptoms and inflammatory markers in women with diarrhea-predominant IBS. Neurogastroenterol Motil. 2017 Jul;29(7). doi: 10.1111/nmo.13037. Epub 2017 Mar 8. PMID 28271623
- [Result] Li B, Liang L, Deng H, Guo J, Shu H, Zhang L. Efficacy and Safety of Probiotics in Irritable Bowel Syndrome: A Systematic Review and Meta-Analysis. Front Pharmacol. 2020 Apr 3;11:332. doi: 10.3389/fphar.2020.00332. eCollection 2020. PMID 32317962
- [Result] Dale HF, Rasmussen SH, Asiller OO, Lied GA. Probiotics in Irritable Bowel Syndrome: An Up-to-Date Systematic Review. Nutrients. 2019 Sep 2;11(9):2048. doi: 10.3390/nu11092048. PMID 31480656
- [Result] Khodadoostan M, Shavakhi A, Sherafat Z, Shavakhi A. Effect of Probiotic Administration Immediately and 1 Month after Colonoscopy in Diarrhea-predominant Irritable Bowel Syndrome Patients. Adv Biomed Res. 2018 Jun 25;7:94. doi: 10.4103/abr.abr_216_17. eCollection 2018. PMID 30050882
- [Result] Niu HL, Xiao JY. The efficacy and safety of probiotics in patients with irritable bowel syndrome: Evidence based on 35 randomized controlled trials. Int J Surg. 2020 Mar;75:116-127. doi: 10.1016/j.ijsu.2020.01.142. Epub 2020 Jan 31. PMID 32014597
- [Result] Gupta A, Khanna S. Fecal Microbiota Transplantation. JAMA. 2017 Jul 4;318(1):102. doi: 10.1001/jama.2017.6466. No abstract available. PMID 28672320
- [Result] Hamazaki M, Sawada T, Yamamura T, Maeda K, Mizutani Y, Ishikawa E, Furune S, Yamamoto K, Ishikawa T, Kakushima N, Furukawa K, Ohno E, Honda T, Kawashima H, Ishigami M, Nakamura M, Fujishiro M. Fecal microbiota transplantation in the treatment of irritable bowel syndrome: a single-center prospective study in Japan. BMC Gastroenterol. 2022 Jul 14;22(1):342. doi: 10.1186/s12876-022-02408-5. PMID 35836115
- [Result] El-Salhy M, Hatlebakk JG, Gilja OH, Brathen Kristoffersen A, Hausken T. Efficacy of faecal microbiota transplantation for patients with irritable bowel syndrome in a randomised, double-blind, placebo-controlled study. Gut. 2020 May;69(5):859-867. doi: 10.1136/gutjnl-2019-319630. Epub 2019 Dec 18. PMID 31852769
- [Result] El-Salhy M, Winkel R, Casen C, Hausken T, Gilja OH, Hatlebakk JG. Efficacy of Fecal Microbiota Transplantation for Patients With Irritable Bowel Syndrome at 3 Years After Transplantation. Gastroenterology. 2022 Oct;163(4):982-994.e14. doi: 10.1053/j.gastro.2022.06.020. Epub 2022 Jun 14. PMID 35709830
- [Result] Xu D, Chen VL, Steiner CA, Berinstein JA, Eswaran S, Waljee AK, Higgins PDR, Owyang C. Efficacy of Fecal Microbiota Transplantation in Irritable Bowel Syndrome: A Systematic Review and Meta-Analysis. Am J Gastroenterol. 2019 Jul;114(7):1043-1050. doi: 10.14309/ajg.0000000000000198. PMID 30908299
- [Result] Bojanova DP, Bordenstein SR. Fecal Transplants: What Is Being Transferred? PLoS Biol. 2016 Jul 12;14(7):e1002503. doi: 10.1371/journal.pbio.1002503. eCollection 2016 Jul. PMID 27404502
- [Result] Francis CY, Morris J, Whorwell PJ. The irritable bowel severity scoring system: a simple method of monitoring irritable bowel syndrome and its progress. Aliment Pharmacol Ther. 1997 Apr;11(2):395-402. doi: 10.1046/j.1365-2036.1997.142318000.x. PMID 9146781
- [Result] Hendriks C, Drent M, Elfferich M, De Vries J. The Fatigue Assessment Scale: quality and availability in sarcoidosis and other diseases. Curr Opin Pulm Med. 2018 Sep;24(5):495-503. doi: 10.1097/MCP.0000000000000496. PMID 29889115
- [Result] Cho HS, Park JM, Lim CH, Cho YK, Lee IS, Kim SW, Choi MG, Chung IS, Chung YK. Anxiety, depression and quality of life in patients with irritable bowel syndrome. Gut Liver. 2011 Mar;5(1):29-36. doi: 10.5009/gnl.2011.5.1.29. Epub 2011 Mar 16. PMID 21461069